CLINICAL TRIAL: NCT04895891
Title: 3D Personalized Modelization of the Hand Using EOS Imaging System
Acronym: M3DME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2019/444
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EOS imaging (Experimental): For each patient, EOS images are compared with computed tomography [CT] images
  Interventions: Device: EOS hand imaging

INTERVENTIONS:
Device: EOS hand imaging — For each patient, EOS images are compared with CT images

SUMMARY:
This study aims to compare the quality of 3D hand modelization with EOS imaging with gold-standard computed tomography

ELIGIBILITY:
Inclusion Criteria:

* Patient with hand/wrist CT required
* Informed consent form signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Data obtained through EOS imaging | Day 60
  Precision and correlation of the 3D modelization of hand is compared between the two imaging methods
Data obtained through standard CT | Day 60
  Precision and correlation of the 3D modelization of hand is compared between the two imaging methods

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No